CLINICAL TRIAL: NCT04218864
Title: Computerized Intervention for Reducing Intimate Partner Violence for Perinatal Women Seeking Mental Health Treatment
Brief Title: Strength for U in Relationship Empowerment
Acronym: SURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Professor of Psychiatry and Human Behavior, Professor of Obstetrics and Gynecology, Professor of Medicine, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 166275; 1R01HD094801-01A1 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2020-01-06 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: IPV; Perinatal; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength for U in Relationship Empowerment (SURE) (Experimental): Theory-driven and derived from empirical support
  Interventions: Behavioral: Strength for U in Relationship Empowerment (SURE)
- Attention, time, and information matched control (Active Comparator): Well-validated
  Interventions: Behavioral: Attention, time, and information matched control

INTERVENTIONS:
Behavioral: Strength for U in Relationship Empowerment (SURE) — A brief computer-based intervention (one session plus one booster session) based on motivational interviewing.
  Arms: Strength for U in Relationship Empowerment (SURE)
Behavioral: Attention, time, and information matched control — A brief computer based intervention (one session plus booster session) that involves viewing of popular television shows
  Arms: Attention, time, and information matched control

SUMMARY:
The objective of this study is to test whether the innovative intervention, "Strength for U in Relationship Empowerment" (SURE), reduces the frequency of IPV more than an attention, time, and information matched control condition in perinatal women seeking mental health care.

DETAILED DESCRIPTION:
Intimate partner victimization (IPV) is a significant social and public health problem among perinatal women. IPV places a woman at high risk for several psychiatric disorders, which transforms the perinatal period from an already challenging process into a potentially overwhelming one. IPV and untreated mental illness during the perinatal period poses a dual risk of adverse physical and emotional outcomes for women and their developing fetus/infant. Given the high rates of IPV among women who seek mental health treatment, mental health clinics compared to other medical settings (e.g. primary care) are more effective sites for focused case finding and intervention. In addition, the presence of IPV increases the likelihood of disengagement from treatment, which could further compromise the health and safety of women and their fetus/infant. Despite the high-risk profile of women with IPV and mental health illness, there are low screening and intervention rates of female mental health patients with IPV within mental health settings.

The objective of this R01 Award is to fill this critical gap by building upon our promising pilot findings to test whether the innovative intervention, "Strength for U in Relationship Empowerment" (SURE), reduces the frequency of IPV more than an attention, time, and information matched control condition in perinatal women seeking mental health care.

The investigators propose a two-group, randomized controlled trial in which 186 perinatal women with IPV women seeking mental health care who will be assigned to either (a) SURE, a computer-delivered, single-session brief intervention plus one interventionist-led phone booster that is consistent with motivational interviewing and informed by the literature on effective interventions for our target population and targeted risk factors, or (b) a computer-delivered control + one interventionist-led phone booster condition. Computer-delivered follow-up assessments will occur at 6 weeks, 3 months, 6 months, and 12 months after the baseline assessment.

Anticipated 25% of planned enrollment recruited by 5/14/2021. Anticipated 50% of planned enrollment recruited by 2/15/2022. Anticipated 75% of planned enrollment recruited by 8/15/2022. Anticipated 100% of planned enrollment recruited by 2/13/2023. Anticipated completion of primary endpoints data analyses by 6/28/2024. Anticipated reporting of results in ClinicalTrials.gov by 6/30/2025.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women
2. Women who have had a baby in the last 12 months
3. Between the ages of 18-45 years old
4. Have reported partner abuse within the last year as measured by the Woman Abuse Screening Tool (WAST)
5. Have sought mental health treatment

Exclusion Criteria:

1. Cannot provide informed consent
2. Unable to understand English
3. No access to the internet or a device with internet access
4. Discomfort with internet use
5. No privacy to view a 40-minute online intervention
6. Screen positive for risk of intimate partner violence that involves severe injury or homicide
7. Screen positive for risk of spyware/stalkerware
8. At one of the two research site, study recruit is unwilling to meet for in-person study visits (if criteria 3-8 are met)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not currently have a plan to share data. However, the team is currently in discussion about sharing data and will update the registration as needed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Started | 65 | 57
Completed | 56 | 50
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control | Total
Number analyzed (Participants) | 65 | 57 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 57 | 122
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 65 | 57 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 53 | 44 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 45 | 33 | 78
  Black | 13 | 16 | 29
  Bi-Racial or Multi-Ethnic | 3 | 3 | 6
  Native American or Native Alaskan | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 57 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 57 | 122
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite Abuse Scale (CAS)
Description: The frequency of IPV will be measured using the Composite Abuse Scale. The Composite Abuse Scale is a 30-item scale with 4 subscales that measure severe combined abuse, emotional abuse, physical abuse, and harassment. Items are scored between 0 and 5, with Never=0 and Daily=5. Scale range is from 0-150. The lower the score, the better or less victimization. Change scores will be used to estimate differences within and between groups.
Time Frame: Baseline, 6-week follow-up, 3, 6, and 12-month follow-up.
Population: All baseline outcome measures were missing for one subject due to a software issue. As a consequence, the outcome analysis was carried out with data from 121 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Number analyzed (Participants) | 64 | 57
units on a scale
  Baseline | 29.13 (20.92) | 27.01 (20.65)
  6-week follow-up | 10.54 (12.02) | 10.02 (12.78)
  3-month follow-up | 9.69 (10.39) | 8.27 (11.06)
  6-month follow-up | 8.89 (12.06) | 8.7 (10.95)
  12-month follow-up | 11.45 (14.56) | 7.5 (12.02)
Statistical Analysis 1: Comparison: Strength for U in Relationship Empowerment (SURE) vs Attention, Time, and Information Matched Control; Linear Mixed regression models (LMM) have been used to identify any difference between the intervention and the control groups over time with regards to the continuous outcomes. Group (intervention vs. control), a 5-category time (baseline, 6 week, 3 month, 6 month, 12 month) and group-by-time interaction are covariates in the model. A random subject intercept is used to account for clustering within subject; Test type: Superiority; p > 0.05, Regression, Linear — Threshold for statistical significance = 0.05; Results presented are unadjusted for any covariates

2. Secondary Outcome: The Positive Affect and Well-being Scale (PAW)
Description: Positive affect and well-being will be measured by using the National Institutes of Health Quality of Life in Neurological Disorders scale for Positive Affect and Well-being a computerized adaptive test 9-item scale. This scale is scored between 1 and 5, with Never=1 and Always=5. Scale range is from 9-45. Higher scores indicate higher positive affect, life satisfaction, or an overall sense of purpose and meaning. Change scores will be used to estimate differences within and between groups.
Time Frame: Baseline, 6-week follow-up, 3, 6, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Number analyzed (Participants) | 64 | 57
units on a scale
  Baseline | 29.39 (7.32) | 29.95 (7.17)
  6-week follow-up | 31.68 (6.43) | 32.05 (6.68)
  3-month follow-up | 33.21 (5.91) | 31.4 (6.84)
  6-month follow-up | 32.64 (6.08) | 30.84 (6.51)
  12-month follow-up | 33.59 (5.75) | 32.93 (6.64)
Statistical Analysis 1: Comparison: Strength for U in Relationship Empowerment (SURE) vs Attention, Time, and Information Matched Control; Statistical analysis strategy is identical to that for the primary outcome; Test type: Superiority; p > 0.05, Regression, Linear — Threshold for statistical significance = 0.05; Results presented are unadjusted for any covariates

3. Secondary Outcome: Perceived Emotional Support (PES)
Description: Perceived emotional support will be measured using a 4-item scale developed by the Patient-Reported Outcomes Measurement Information System . Patient-Reported Outcomes Measurement Information System is a National Institutes of Health Roadmap initiative that provides precise, reliable, valid, and standardized questionnaires measuring patient-reported outcomes across the domains of physical, mental, and social health. The Patient-Reported Outcomes Measurement Information System .Emotional Support item bank specifically aims to measure perceived feelings of being cared for and valued as a person. This scale is scored between 1 and 5, with Never=1 and Always=5. Scale range is from 4-20. A higher Patient-Reported Outcomes Measurement Information System score represents increased emotional support. Change scores will be used to estimate differences within and between groups.
Time Frame: Baseline, 6-week follow-up, 3, 6, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Number analyzed (Participants) | 64 | 57
units on a scale
  Baseline | 14.61 (4.15) | 14.89 (4.16)
  6- Week | 15.41 (3.63) | 15.32 (4.23)
  3- Month | 15.75 (3.45) | 14.77 (4.46)
  6- Month | 15.15 (3.54) | 15.12 (3.49)
  12-Month | 16.02 (3.67) | 15.58 (4)
Statistical Analysis 1: Comparison: Strength for U in Relationship Empowerment (SURE) vs Attention, Time, and Information Matched Control; Statistical analysis strategy is identical to that for the primary outcome; Test type: Superiority; p > 0.05, Regression, Linear — Threshold for statistical significance = 0.05; Results presented are unadjusted for any covariates

4. Other Pre Specified Outcome: Personal Progress Scale-Revised (PPS-R)
Description: Empowerment will be measured using the Personal Progress Scale-Revised for measuring skills, social supports, and resources to cope more effectively with relationship stress and trauma. The Personal Progress Scale-Revised is a 28-item scale scored between 1 and 7, with 1=Almost Never and 7=Almost Always. Scale range is from 28-196. Higher scores indicating higher empowerment. Change scores will be used to estimate differences within and between groups.
Time Frame: Baseline, 6-week follow-up, 3, 6, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Number analyzed (Participants) | 64 | 57
units on a scale
  Baseline | 129.53 (21.66) | 132.56 (22.62)
  6-Week | 109.08 (14.39) | 113.66 (11.72)
  3-Month | 111.4 (13.4) | 113.74 (14.11)
  6-Month | 111.42 (14.01) | 113.84 (14.11)
  12-Month | 114.1 (16.44) | 110.87 (12.03)
Statistical Analysis 1: Comparison: Strength for U in Relationship Empowerment (SURE) vs Attention, Time, and Information Matched Control; Statistical analysis strategy is identical to that for primary outcome; Test type: Superiority; p > 0.05, Regression, Linear — Threshold for statistical significance = 0.05; Results presented are unadjusted for any covariates

5. Other Pre Specified Outcome: Self-efficacy (GSE)
Description: Self-efficacy will be measured using the General Self-Efficacy Scale a 10-item self-report measure. It measures personal competence to deal effectively with a variety of stressful situations. The General Self-Efficacy Scale is scored from 10-40, with 1=Not at all true and 4=Exactly true. A higher score indicates more self-efficacy. Change scores will be used to estimate differences within and between groups.
Time Frame: Baseline, 6-week follow-up, 3, 6, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
Number analyzed (Participants) | 64 | 57
units on a scale
  Baseline | 28.45 (4.57) | 27.34 (4.8)
  6- Week | 28.71 (4.17) | 28.68 (5.23)
  3- Month | 29.67 (3.82) | 29.57 (5.32)
  6- Month | 29.49 (4.23) | 28.84 (4.58)
  12-Month | 30.72 (3.94) | 29.79 (4.7)
Statistical Analysis 1: Comparison: Strength for U in Relationship Empowerment (SURE) vs Attention, Time, and Information Matched Control; Statistical Analysis strategy is identical to that for primary outcome measure; Test type: Superiority; p > 0.05, Regression, Linear — Threshold for statistical significance = 0.05; Results presented are unadjusted for any covariates

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 6-weeks, 3-months, 6 months , and 12-months after baseline assessment
Description: Systematic assessment: The study research staff conducted a standard structured interview at each follow-up period. Specific pregnancy-related medical conditions resulting in hospitalization were not evaluated.
Arm/Group | Strength for U in Relationship Empowerment (SURE) | Attention, Time, and Information Matched Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/57
Serious Adverse Events (participants affected / at risk) | 24/65 | 17/57
Other Adverse Events (participants affected / at risk) | 0/65 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength for U in Relationship Empowerment (SURE) (N=65) | Attention, Time, and Information Matched Control (N=57)
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) — Specific events include hospitalizations due to stillbirth, shortened cervix, and pregnancy-related psoriasis and pulmonary edema.
Hospitalization (Renal and urinary disorders) | 2 (2) | 1 (1) — Specific events include hospitalizations due to gallbladder removal and kidney infection.
IPV Altercation (non-study related) (Social circumstances) | 15 (37) | 9 (19) — All non-study related.
Hospitalization (Psychiatric disorders) | 2 (3) | 4 (4) — Specific events include hospitalizations for depression, stress and past trauma, suicidal ideation and/or attempt, generic mental health reasons, and not feeling safe at home in terms of self-harm.
Housing (Social circumstances) | 1 (1) | 1 (1) — Specific events include danger or threats from someone other than an intimate partner and being in the vicinity of gunshots during a neighborhood dispute.
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Specific event was a hospitalization due to a pelvic infection.
Hospitalization (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Specific event was a hospitalization due to ear pain and vertigo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT04218864/Prot_SAP_000.pdf